CLINICAL TRIAL: NCT06140264
Title: Short Term Effect of Acupuncture Dry Needle in Treatment of Chronic Mechanical Low Back Pain: A Randomized Controlled Clinical Trial
Brief Title: Effect of Acupuncture Dry Needle in Treatment of Chronic Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/022/035
Record Dates: First submitted 2023-07-09; First posted 2023-11-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain
Keywords: Acupuncture dry needle; Chronic mechanical low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture dry needle (Active Comparator): This group received acupuncture dry needle over trigger points of back muscles followed by stretching and strengthening exercises for back muscles, 2 sessions per week for 2 weeks.
  Interventions: Other: Acupuncture dry needle
- Stretching and strengthening exercises (No Intervention): This group received only stretching and strengthening exercises for back muscles.

INTERVENTIONS:
Other: Acupuncture dry needle — The muscles that have been treated iliocostalis lumborum, quadratus lumborum, gluteus medius and piriformis muscles. The patients received 2 sessions per week for 2 weeks.
  Arms: Acupuncture dry needle

SUMMARY:
Low back pain affects about 60% to 90% of the working-age population in modern industrial society. Chronic mechanical low back pain (CMLBP) is the most common problem of the working-age population in modern industrial society; it causes a substantial economic burden due to the wide use of medical services and absence from work. The purpose of this trial was to evaluate the short-term effect of acupuncture dry needle in treatment of chronic mechanical low back pain.

DETAILED DESCRIPTION:
Low back pain affects about 60% to 90% of the working-age population in modern industrial society. Chronic mechanical low back pain (CMLBP) is the most common problem of the working-age population in modern industrial society; it causes a substantial economic burden due to the wide use of medical services and absence from work. The purpose of this trial was to evaluate the short-term effect of acupuncture dry needle in treatment of chronic mechanical low back pain. Thirty patients their age ranged from 20 - 45 years participated in our study and divided randomly into two equal groups suffering from nonspecific low back pain. The first group (A) consist of 15 patients receiving acupuncture dry needle over trigger points of back muscles followed by stretching and strengthening exercises for back muscles, the second group (B) consist of 15 patients receiving only stretching and strengthening exercises for back muscles. The following parameters including pain severity, functional disability and lumbar range of motion (flexion, extension, right side bending and left side bending) were measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from 20 to 45 years old.
2. Pain of at least 30 mm to 70 mm on a visual analogue scale (VAS) from 0 mm (no pain) to 100 mm (worst imaginable pain).
3. Presence of MTrPs at least in 4 muscles on any side.
4. Patients had lower back myofascial pain syndrome for at least 3 months ago.

Exclusion Criteria:

A history of previous back surgery, neurologic deficit, current lower extremity symptoms, cardiopulmonary disease with decreased activity tolerance, rheumatologic conditions, polyarticular osteoarthritis, rheumatoid arthritis and advanced lumbar degenerative disease, patients receiving other treatment in the form of physical therapy or medication for the duration of the study that may interfere with the results of this study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Four weeks
  Pain was assessed by Visual Analog Scale (VAS). VAS is a scale that allows continuous data analysis and uses a 10 cm line with 0 in one end (no pain) and 10 (worst pain) on the other end. Patients were asked to place a mark along the line to denote their level of pain.

SECONDARY OUTCOMES:
Functional disability | Four weeks
  Functional disability of each patient was assessed by Oswestery disability questionnaire. It is valid and reliable tool. It is consists of 10 multiple choice questions for back pain, patient select one sentence out of six that best describe his pain, Higher scores indicated great pain. Scores (0-20%) minimal disability, Scores (20%- 40%) moderate, Scores (40% - 60%) severe, Scores (60%-80%) crippled, Scores (80% - 100%) patients are confined to bed.
Lumbar range of motion | Four weeks
  Modified-modified Schober flexion technique was used based on the work of Williams et al. This method is reliable and valid in measuring range of motion of lumbar flexion. The investigator stood behind the standing patient to identify the posterior superior iliac spines with her or his thumbs, and then an ink mark was drawn along the midline of the lumbar spine horizontal to the posterior superior iliac spines. Another ink mark was made 15 cm above the original mark; the distance between superior and inferior skin marks was measured. Then the investigator instructed the patient to bend forward into full lumbar flexion and the new distance between superior and inferior skin marks was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Walid Kamal Abdelbasset, Al Kharj, Riyadh Region, Saudi Arabia